CLINICAL TRIAL: NCT02091336
Title: Oral Antidiabetic Agents on Gestational Diabetes: Modulating Effect on Fetal Growth - a Clinical Randomized Trial
Brief Title: Oral Antidiabetic Agents in Pregnancy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OAGM-001
Record Dates: First submitted 2014-02-25; First posted 2014-03-19 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-01

CONDITIONS: Gestational Diabetes
Keywords: gestational diabetes; metformin; glyburide; fetal growth; capillar glucose
MeSH Terms: conditions — Diabetes, Gestational | interventions — Metformin; Glyburide; Glucovance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glyburide (Active Comparator): Glyburide 2,5 mg
  Interventions: Drug: Glyburide
- Metformin (Active Comparator): Metformin 500mg bid
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — patients treatment
  Other Names: Glucophage, Glifage
  Arms: Metformin
Drug: Glyburide — patients treatment
  Other Names: Glibenclamida, Glucovance
  Arms: Glyburide

SUMMARY:
The aim of this study is to determine the efficacy of oral treatment with glyburide and metformin controlling excessive fetal growth in women with gestational diabetes, using insulin as a ransom on no response to oral treatment .

It is randomized with women who seek care at the Outpatient Diabetes in Pregnancy in our hospital trial Eligible women between 18 - 45anos diagnosed with gestational diabetes , according to the WHO criteria , ratified the public network for prenatal care at the Clinic for Diabetes and Pregnancy HCPA .

Women with singleton pregnancy and gestational age not exceeding 30 weeks at the time of enrollment.

Pregnant women with indication for pharmacological treatment will be invited to randomization to use of oral , glyburide or metformin antidiabetic .

At regular intervals of 2 - 3 weeks fetal growth will be measured with obstetric ultrasonography , until birth.

The primary outcomes will be :

( 1 ) weight and gestational age at birth and the index of large for gestational age fetuses ( ≥ 90th percentile for gestational age ) ( 2 ) the use of insulin to achieve glycemic targets according to fetal growth , as an indirect measure of the inefficiency of oral medications .

DETAILED DESCRIPTION:
The procedures for monitoring metabolic and obstetrical control , assessments of fetal well -being and indications for interruption are usually adopted in the Outpatient Diabetes and Pregnancy of the institution.

- Patients will be followed since their first appointment in our hospital, around the 20th week of pregnancy- until 8 weeks after labor and delivery. That being said, patients will be followed by an average of 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Eligible women between 18-45 years diagnosed with gestational diabetes, according to the WHO criteria (19), ratified the public network for prenatal care at the Clinic for Diabetes and Pregnancy.
* Women with singleton pregnancy and gestational age not exceeding 30 weeks at the time of enrollment, calculated from ultrasound (U.S.) Obstetric performed before the 20th week of pregnancy will be enrolled.

Exclusion Criteria:

* Women who present enrollment in the diagnosis of chronic hypertension, heart disease or chronic lung disease intrauterine restricted or preterm labor, growth, or even chronic diarrhea will be excluded

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
fetal growth | up to 9 months
  fetal growth will be assessed every 3 weeks by obstetric ultrasound during pregnancy until delivery

SECONDARY OUTCOMES:
insulin requirements to achieve glucose targets | up to 9 months
  every week patients will have one whole day in the hospital to monitor capillar glucose levels

OTHER OUTCOMES:
hypoglycaemia | up to 9 months
  medications will be suspended if patients present with repeated hypoglycaemia
maternal weight gain | up to 9 months
neonatal 5th minute apgar | 5 minutes after birth
neonatal hypoglycaemia and respiratory distress | 48 hours after birth
neonatal need of intensive care | 48 hours after birth
need of c section | day of birth

CONTACTS AND LOCATIONS:
Overall Officials: Maria Lucia R Oppermann, PhD Prf, Study Chair — HCPA-UFRGS; Vanessa K Genro, PhD, Principal Investigator — HCPA
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil